CLINICAL TRIAL: NCT01587573
Title: Pivotal Validation Study of Salivary Biomarkers for the Risk Stratification of Patients With Lesions Suspicious for Oral Squamous Cell Carcinoma
Brief Title: Developing an In-vitro Diagnostic Risk-Stratification Test for Oral Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PeriRx (Industry)
Responsible Party: Sponsor
Other Study IDs: PeriRx-1
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-05

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: salivary biomarkers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell free saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- oral lesions: oral lesions suspicious for squamous cell carcinoma with saliva collection prior to clinically driven oral biopsy
  Interventions: Other: saliva collection prior to clinically driven oral biopsy

INTERVENTIONS:
Other: saliva collection prior to clinically driven oral biopsy — cell free saliva to be used to measure mRNA and proteins by PCR and ELISA

SUMMARY:
The purpose of this study is to verify the discriminatory value of previously identified salivary transcriptome and proteome markers for oral squamous cell cancer in an intended use population of patients with oral lesions suspicious for cancer.

DETAILED DESCRIPTION:
Saliva samples are collected from patients before clinically driven oral biopsy for lesions suspicious for cancer. Specimens are processed by laboratory personnel blinded to the tissue diagnosis. Six pre-specified mRNA markers (IL1b, IL8, SAT, DUSP1, OAZ1 and S100P) are measured by polymerase chain reaction. Markers are compared in cancer and control by raw Ct values as well as by delta Ct after adjustment for housekeeping gens. Appropriate housekeeping genes are identified in a random subset of cancer and control patients and then verified in the remaining subjects. Predictive models are generated by a pre-specified method and robustness evaluated by bootstrap analysis. The model is then further validated in a second cohort. Three pre-specified protein markers (IL8, IL1B, and M2BP) are a secondary endpoint and will also be compared in cancer and control patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for biopsy of an oral lesion suspicious for squamous cell cancer

Exclusion Criteria:

* Patients with known prior oral malignancy in last 2 years or other cancer in last 5 years other than non melanoma skin cancer or with immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with oral lesions suspicious for squamous cell cancer and scheduled for clinically driven biopsy
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2012-04 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Test specificity at 90% sensitivity | at study completion as well as after model development following enrollment of the first 30 patents with cancer
  Based on multimarker test score

SECONDARY OUTCOMES:
Validation of individual mRNA and protein markers | After enrollment of 30 patients with cancer
  Based on comparison of cancer and controls
Validation of a pre-specified multi marker model | After enrollment of 30 patients with cancer
  Based on combined sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Jack L Martin, MD, Principal Investigator — PeriRx, LLC; Marc Surkin, MD, Study Chair — Main Line Health System
Locations (5):
- United States (5):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Department of Surgery, Michigan Sate University, East Lansing, Michigan
  - St. John Providence Health System, Warren, Michigan
  - Main Line Health System, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martin JL. Validation of Reference Genes for Oral Cancer Detection Panels in a Prospective Blinded Cohort. PLoS One. 2016 Jul 13;11(7):e0158462. doi: 10.1371/journal.pone.0158462. eCollection 2016. PMID 27411053